CLINICAL TRIAL: NCT06769334
Title: Digital Health Intervention to Improve Neurodevelopmental Outcomes for Young Childhood Cancer Survivors in Underserved Communities
Brief Title: Preparing for Life and Academics for Young Childhood Cancer Survivors
Acronym: PLAY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Emily Moscato, Principal Investigator, Nationwide Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00004302; K08CA290060 (NIH)
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Childhood Cancer
Keywords: positive parenting; development; school readiness; digital health; caregiver stress; school advocacy
MeSH Terms: conditions — Neoplasms; Caregiver Burden

STUDY DESIGN:
Masking Description: Staff members who are completing the coding for the standardized parent-child interaction task will be blinded to time point.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preparing for Life and Academics for Young (PLAY) survivors program (Experimental): PLAY is a digital health intervention involving 7 self-directed web-modules and up to 10 virtual coaching sessions conducted weekly to biweekly (7 paired plus up to 3 booster sessions) for caregivers of young childhood cancer survivors (3-6 years). The module content focuses on psychoeducation and positive parenting skills and the coaching focuses on live practice of positive parenting skills.
  Interventions: Other: PLAY Program

INTERVENTIONS:
Other: PLAY Program — The PLAY Program is a web-based program created for caregivers of childhood cancer survivors. The program consists of seven modules with the following topics: 1) Introduction to the program 2) Self-Care 3) Relationships 4) Getting Ready for School 5) Talking, Reading, and Counting together 6) Social and Emotional Development 7) Review Module. The program is meant to be completed over approximately three months, and caregivers in the program will meet with a coach on a weekly or bi-weekly basis to discuss what they learned in the modules and how to practice it in their daily lives.

SUMMARY:
The goal of this clinical trial is to test and improve an online program for caregivers of young childhood cancer survivors called the Preparing for Life and Academics for Young Survivors program (PLAY). The PLAY program was created with a group of caregivers of young children with cancer and healthcare providers. Ultimately, investigators hope to see if the program can improve positive parenting behaviors, reduce caregiver stress, and help get young children ready for school. In the preliminary phase of this clinical trial, investigators are aiming to answer these questions:

1. Are caregivers of childhood cancer survivors willing to participate in the PLAY program and complete assessments before and after the program?
2. Do caregivers of childhood cancer survivors rate the PLAY program as easy to use?
3. Are caregivers of childhood cancer survivors satisfied with the PLAY program?
4. How can the PLAY program be improved in the future?
5. Does PLAY help improve how caregivers interact and read with their children or how they manage their own stress?

When the child is transitioning to maintenance phase therapies or is no longer actively in cancer treatment, caregivers will be invited to participate. If they agree to participate, they will complete surveys when they begin the study as well as a videotaped interaction task reading and playing with their child. Children will complete brief developmental testing at the beginning of the program.

Caregivers will then complete the PLAY Program, which will involve completing 7 weekly or bi-weekly online modules and meeting with a trained coach by videoconference for up to 10 one-hour sessions over three months. Sessions will focus on helping their child get ready for school and helping their family adjust and cope with stress.

Caregivers will repeat the surveys and videotaped interaction task again three months later, after the PLAY program is completed. They will also be invited to participate in an interview to learn about their experience in the program.

This study will happen over two phases. Participants in Phase I of this study will complete all parts of the study as described above. Participants in Phase II (beginning in winter 2025) will complete all parts of the study as described above and a six month follow up that will involve repeating the similar questionnaires and an additional videotaped interaction with their child. Teachers of children will also take part in Phase II with questionnaires at baseline and 3-months later, after participants have completed the PLAY program.

DETAILED DESCRIPTION:
This study will occur in two phases. Phase I will involve rapid cycle testing of the intervention and Phase II will be a single-arm trial of the PLAY program.

For phase I, the aim of this study is to refine PLAY to optimize feasibility and acceptability (ORBIT Phase Ib) through rapid-cycle testing with families of YCCS (n=5 per group, up to 15 total) in partnership with advisory boards comprised of 10 families of YCCS, including rural and Appalachian YCCS, and 10 healthcare providers ("co-designers"). Rapid cycle testing to iteratively refine PLAY will determine its optimal timing, dose, and duration until three caregivers sequentially endorse above-average usability (System Usability Scale score >68), feasibility, and acceptability ratings (>80%), or up to n=15 families have completed the PLAY program.

Following rapid cycle testing, phase II will involve a single-arm trial of PLAY program with up to 20 new families of YCCS to evaluate the refined program's feasibility, acceptability, and proof-of-concept. Caregivers will be recruited and will participate using analogous procedures and measures, as described in Phase I, with the addition of 6-month post-baseline assessments.

ELIGIBILITY:
For the caregiver:

* Caregiver is the legal guardian of the child (e.g., mothers, fathers, grandparents, adoptive parents)
* Caregiver lives with the child more than 50% of the time
* Caregiver primary language is English
* Caregiver lives within 150 miles of Nationwide Children's Hospital

For the childhood cancer survivor:

* Received treatment for their cancer (e.g., chemotherapy, surgical resection, radiation therapy)
* Completed cancer treatment or on maintenance therapy only, without evidence of recurrent disease
* Childhood cancer survivor is currently between the ages of 3 years old to 6 years old, but no older than 6.5 years old at study enrollment

Exclusion Criteria for the childhood cancer survivor:

* Has a documented neurodevelopmental disorder prior to their cancer diagnosis (e.g., neurofibromatosis, tuberous sclerosis, Down's syndrome, autism)
* Did not receive any treatment for their cancer (e.g., chemotherapy, surgical resection, radiation)
* Treated for a benign tumor

For the teacher:

Classroom or daycare teacher of the childhood cancer survivor

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
System Usability Scale | 3 months post-enrollment
  This is a 10-item measure that will quantitatively assess usability of our web-based program. The SUS measures how accessible the website is and whether participants can understand the content of the website on a scale of 0-100. We will continue to recruit until our website has achieved an average score of >68% (above average).
Intervention Appropriateness Measure (IAM) | 3 Months Post-Enrollment
  Participants will use this four-item measure to rate the appropriateness of the PLAY program. Each item is rated from 1-5 and the final score for the measure is the average number for all answers. A higher score means a participant rated the PLAY program as more appropriate, an overall score of 4 or higher (80%) means a participant found the program to be appropriate.
Acceptability of Intervention Measure (AIM) | 3 Months Post-Enrollment
  This is a four-item measure that will have participants rate the acceptability of the PLAY program. Each item is rated from 1-5 and the final score for the measure is the average number for all answers. A higher score means a participant rated the PLAY program as more acceptable, an overall score of 4 or higher (80%) means a participant found the program to be acceptable.
Adapted Website Evaluation Questionnaire (WEQ) | 3 months post-enrollment
  This measure will assess accessibility and satisfaction with the PLAY Program. Four overall items will be rated from 1-10 by participants. The overall score will be the average response across items. A higher score indicates higher satisfaction with the program. Overall scores of 8 or higher (> 80%) are an indication of satisfaction with the PLAY program.
Feasibility of the PLAY program | 3 month post-enrollment (Phase I); 3 and 6 month post-enrollment (Phase II)
  Enrollment rate (#enrolled/#approached; milestone greater than or equal to 50%), completion rate (# completing core PLAY sessions/#enrolled; milestone greater than or equal to 75%), retention rate (#completers of 3 and 6 month assessments/ # enrolled at baseline; milestone greater than or equal to 70%); Caregivers who rate the intervention greater than or equal to 80% on the Feasibility Intervention Measure (FIM; milestone >80%), which is a four-item measure. Each item is rated from 1-5 and the final score for the measure is the average number for all answers. A higher score means a participant rated the PLAY program as more feasible, an overall score of 4 or higher (80%) means a participant found the program to be feasible.

SECONDARY OUTCOMES:
Play and Alternative Learning Strategies parent-child interaction coding | Baseline, 3 and 6 month follow up (Phase II)
  Caregivers will record themselves playing with with their child for at least 10 minutes for a measure of observed positive parenting behaviors which will be rated with the standardized Play and Learning Strategies coding scheme by trained raters blinded to timepoint. The coding scheme involves 1 to 5 Likert scale ratings of positive parenting behaviors (i.e., warmth, contingent responsiveness, maintaining, verbal scaffolding, demonstration/physical teaching). Proof of concept will be determined if 8 of 15 caregivers demonstrate improvements by greater than 1 point on observed positive parenting behaviors from baseline.
Parenting Stress Index-Short Form | Baseline, 3 and 6 months post-enrollment (Phase II)
  Caregivers will complete the Parenting Stress Inventory, Short Form (PSI-SF), yielding a Total Parenting Stress Score. Proof-of-concept will be determined if at least 8 of 15 caregivers report either maintenance of non-clinical levels of parenting stress or reduction to non-clinical levels post-intervention (i.e., Total Parenting Stress < 85th percentile).
Hospital Depression and Anxiety Scale (HADS) | Baseline, 3 and 6 months post-enrollment (Phase II)
  Caregivers will complete the Hospital Anxiety and Depression Scale (HADS) which yields Anxiety and Depression Total Scores. Proof-of-concept will be determined if at least 8 of 15 caregivers report either maintenance of non-clinical levels of anxiety/depression or reduction to non-clinical levels post-intervention (i.e., HADS scores less than a score of 8).

OTHER OUTCOMES:
Behavior Rating Inventory of Executive Function (BRIEF-P or -2) | Baseline, 3 and 6 months post-enrollment (Phase II)
  Caregivers and teachers will complete the Behavior Rating Inventory of Executive Function, Preschool (BRIEF-P; ages 2 to 5 years) or the BRIEF-2 (ages 5 years+), yielding a General Executive Composite. Proof of concept will be determined if 8 of 15 caregivers and teachers report either that the child has maintained non-clinical levels of executive functioning problems or has reduced executive functioning problems to the non-clinical range post-intervention (i.e., General Executive Composite T-score less than or equal to 65).
Adaptive Behavior Assessment System, Third Edition (ABAS-3; Pre-Academics or Functional Academics subscale) | Baseline, 3 and 6 months post-enrollment (Phase II)
  Caregivers and teachers will also complete the Adaptive Behavior Assessment System, Third Edition (ABAS-3; Pre-Academics or Functional Academics subscale). Proof of concept will be determined if 8 of 15 caregivers and teachers either report that the child has maintained on track performance for pre-academic skills, or has improved in their pre-academic skills to a non-delayed range (i.e., scaled score greater than or equal to 6).

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected, deidentified quantitative IPD for the primary and secondary outcomes of the study for participants who consent to have their data shared.
Supporting Information: Study Protocol
Time Frame: IPD will be made available after the primary outcomes manuscript is published and will be available for at least seven years post study-closure.
Access Criteria: Interested parties will be able to access the IPD by contacting the PI or through request at the Inter-university Consortium for Political and Social Research.

REFERENCES:
- [Background] Moscato EL, Darow E, Quach J, M Winning A, Schmidt M, Wade SL, Gerhardt CA, Sezgin E. Usability Testing of an Internet-Based Responsive Parenting Program for Caregivers of Young Survivors of Childhood Cancer Living in Rural and Appalachian Communities: Mixed Methods Study. JMIR Pediatr Parent. 2025 Aug 5;8:e70055. doi: 10.2196/70055. PMID 40764035
- [Background] Yao N, Alcala HE, Anderson R, Balkrishnan R. Cancer Disparities in Rural Appalachia: Incidence, Early Detection, and Survivorship. J Rural Health. 2017 Sep;33(4):375-381. doi: 10.1111/jrh.12213. Epub 2016 Sep 7. PMID 27602545
- [Background] Wochos GC, Semerjian CH, Walsh KS. Differences in parent and teacher rating of everyday executive function in pediatric brain tumor survivors. Clin Neuropsychol. 2014;28(8):1243-57. doi: 10.1080/13854046.2014.971875. Epub 2014 Oct 24. PMID 25343533
- [Background] Winter AL, Conklin HM, Tyc VL, Stancel H, Hinds PS, Hudson MM, Kahalley LS. Executive function late effects in survivors of pediatric brain tumors and acute lymphoblastic leukemia. J Clin Exp Neuropsychol. 2014;36(8):818-30. doi: 10.1080/13803395.2014.943695. Epub 2014 Aug 15. PMID 25126830
- [Background] Willard VW, Qaddoumi I, Zhang H, Huang L, Russell KM, Brennan R, Wilson MW, Rodriguez-Galindo C, Phipps S. A longitudinal investigation of parenting stress in caregivers of children with retinoblastoma. Pediatr Blood Cancer. 2017 Apr;64(4):10.1002/pbc.26279. doi: 10.1002/pbc.26279. Epub 2016 Nov 3. PMID 27808461
- [Background] Willard VW, Gordon ML, Means B, Brennan RC, Conklin HM, Merchant TE, Vinitsky A, Harman JL. Social-Emotional Functioning in Preschool-Aged Children With Cancer: Comparisons Between Children With Brain and Non-CNS Solid Tumors. J Pediatr Psychol. 2021 Aug 11;46(7):790-800. doi: 10.1093/jpepsy/jsab018. PMID 33682007
- [Background] Willard VW, Cox LE, Russell KM, Kenney A, Jurbergs N, Molnar AE Jr, Harman JL. Cognitive and Psychosocial Functioning of Preschool-Aged Children with Cancer. J Dev Behav Pediatr. 2017 Oct;38(8):638-645. doi: 10.1097/DBP.0000000000000512. PMID 28937451
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Ward R, Reynolds JE, Pieterse B, Elliott C, Boyd R, Miller L. Utilisation of coaching practices in early interventions in children at risk of developmental disability/delay: a systematic review. Disabil Rehabil. 2020 Oct;42(20):2846-2867. doi: 10.1080/09638288.2019.1581846. Epub 2019 Apr 25. PMID 31021669
- [Background] Wade SL, Cassedy AE, Shultz EL, Zang H, Zhang N, Kirkwood MW, Stancin T, Yeates KO, Taylor HG. Randomized Clinical Trial of Online Parent Training for Behavior Problems After Early Brain Injury. J Am Acad Child Adolesc Psychiatry. 2017 Nov;56(11):930-939.e2. doi: 10.1016/j.jaac.2017.09.413. Epub 2017 Sep 14. PMID 29096775
- [Background] Vance YH, Eiser C. The school experience of the child with cancer. Child Care Health Dev. 2002 Jan;28(1):5-19. doi: 10.1046/j.1365-2214.2002.00227.x. PMID 11856182
- [Background] Van Schoors M, Caes L, Knoble NB, Goubert L, Verhofstadt LL, Alderfer MA; Guest Editors: Cynthia A. Gerhardt, Cynthia A. Berg, Deborah J. Wiebe and Grayson N. Holmbeck. Systematic Review: Associations Between Family Functioning and Child Adjustment After Pediatric Cancer Diagnosis: A Meta-Analysis. J Pediatr Psychol. 2017 Jan 1;42(1):6-18. doi: 10.1093/jpepsy/jsw070. PMID 28173163
- [Background] Snaith RP. The Hospital Anxiety And Depression Scale. Health Qual Life Outcomes. 2003 Aug 1;1:29. doi: 10.1186/1477-7525-1-29. PMID 12914662
- [Background] Schorr E, Wade SL, Taylor HG, Stancin T, Yeates KO. Parenting styles as a predictor of long-term psychosocial outcomes after traumatic brain injury (TBI) in early childhood. Disabil Rehabil. 2020 Aug;42(17):2437-2443. doi: 10.1080/09638288.2019.1602676. Epub 2019 Apr 21. PMID 31006276
- [Background] Rodriguez EM, Dunn MJ, Zuckerman T, Vannatta K, Gerhardt CA, Compas BE. Cancer-related sources of stress for children with cancer and their parents. J Pediatr Psychol. 2012 Mar;37(2):185-97. doi: 10.1093/jpepsy/jsr054. Epub 2011 Aug 13. PMID 21841187
- [Background] Robinson KE, Kuttesch JF, Champion JE, Andreotti CF, Hipp DW, Bettis A, Barnwell A, Compas BE. A quantitative meta-analysis of neurocognitive sequelae in survivors of pediatric brain tumors. Pediatr Blood Cancer. 2010 Sep;55(3):525-31. doi: 10.1002/pbc.22568. PMID 20658625
- [Background] Riggs NR, Jahromi LB, Razza RP, Dillworth-Bart JE, Mueller U. Executive function and the promotion of social-emotional competence. Journal of Applied Developmental Psychology. 2006;27(4):300-9.
- [Background] Potter JL, Wade SL, Walz NC, Cassedy A, Stevens MH, Yeates KO, Taylor HG. Parenting style is related to executive dysfunction after brain injury in children. Rehabil Psychol. 2011 Nov;56(4):351-8. doi: 10.1037/a0025445. Epub 2011 Sep 19. PMID 21928918
- [Background] Phillips SM, Padgett LS, Leisenring WM, Stratton KK, Bishop K, Krull KR, Alfano CM, Gibson TM, de Moor JS, Hartigan DB, Armstrong GT, Robison LL, Rowland JH, Oeffinger KC, Mariotto AB. Survivors of childhood cancer in the United States: prevalence and burden of morbidity. Cancer Epidemiol Biomarkers Prev. 2015 Apr;24(4):653-63. doi: 10.1158/1055-9965.EPI-14-1418. PMID 25834148
- [Background] Peterson CC, Drotar D. Family impact of neurodevelopmental late effects in survivors of pediatric cancer: review of research, clinical evidence, and future directions. Clin Child Psychol Psychiatry. 2006 Jul;11(3):349-66. doi: 10.1177/1359104506064980. PMID 17080773
- [Background] Patel SK, Wong AL, Cuevas M, Van Horn H. Parenting stress and neurocognitive late effects in childhood cancer survivors. Psychooncology. 2013 Aug;22(8):1774-82. doi: 10.1002/pon.3213. Epub 2012 Oct 25. PMID 23097416
- [Background] Owens JA, Spirito A, McGuinn M. The Children's Sleep Habits Questionnaire (CSHQ): psychometric properties of a survey instrument for school-aged children. Sleep. 2000 Dec 15;23(8):1043-51. PMID 11145319
- [Background] Ostrom QT, Gittleman H, Xu J, Kromer C, Wolinsky Y, Kruchko C, Barnholtz-Sloan JS. CBTRUS Statistical Report: Primary Brain and Other Central Nervous System Tumors Diagnosed in the United States in 2009-2013. Neuro Oncol. 2016 Oct 1;18(suppl_5):v1-v75. doi: 10.1093/neuonc/now207. No abstract available. PMID 28475809
- [Background] Neu MA, Schlecht J, Schmidt MF, Robinson AL, Spix C, Grabow D, Kaatsch P, Erdmann F, Faber J, Urschitz MS; IkidS Study Group. Mental health and health-related quality of life in preschool-aged childhood cancer survivors. Results of the prospective cohort study ikidS-OEVA. Pediatr Blood Cancer. 2021 Aug;68(8):e29039. doi: 10.1002/pbc.29039. Epub 2021 May 7. PMID 33960635
- [Background] Moscato E, Patronick J, Wade SL. Family functioning and adaptation following pediatric brain tumor: A systematic review. Pediatr Blood Cancer. 2022 Feb;69(2):e29470. doi: 10.1002/pbc.29470. Epub 2021 Nov 29. PMID 34842339
- [Background] McKercher KA. Beyond Sticky Design: Codesign for Real Inscope Books; 2020.
- [Background] McClelland MM, Acock AC, Morrison FJ. The impact of kindergarten learning-related skills on academic trajectories at the end of elementary school. Early childhood research quarterly. 2006;21(4):471-90.
- [Background] Merz EC, Landry SH, Montroy JJ, Williams JM. Bidirectional Associations Between Parental Responsiveness and Executive Function During Early Childhood. Soc Dev. 2017 Aug;26(3):591-609. doi: 10.1111/sode.12204. Epub 2016 Jul 22. PMID 28860682
- [Background] Maurice-Stam H, Oort FJ, Last BF, Brons PP, Caron HN, Grootenhuis MA. Longitudinal assessment of health-related quality of life in preschool children with non-CNS cancer after the end of successful treatment. Pediatr Blood Cancer. 2008 May;50(5):1047-51. doi: 10.1002/pbc.21374. PMID 17914734
- [Background] Mann TD, Hund AM, Hesson-McInnis MS, Roman ZJ. Pathways to school readiness: Executive functioning predicts academic and social-emotional aspects of school readiness. Mind, Brain, and Education. 2017;11(1):21-31.
- [Background] Maggard BL, Gies LM, Sidol CA, Moscato EL, Schmidt M, Landry SH, Makoroff KL, Rhine TD, Wade SL. Online Intervention for Caregivers of Children with Early Traumatic Brain Injury: Pilot Trial. J Pediatr Psychol. 2023 Mar 20;48(3):205-215. doi: 10.1093/jpepsy/jsac080. PMID 36240452
- [Background] Loyd BH, Abidin RR. Revision of the Parenting Stress Index. J Pediatr Psychol. 1985 Jun;10(2):169-77. doi: 10.1093/jpepsy/10.2.169. No abstract available. PMID 4020601
- [Background] Lansford JE, Odgers CL, Bradley RH, Godwin J, Copeland WE, Rothenberg WA, Dodge KA. The HOME-21: A revised measure of the home environment for the 21st century tested in two independent samples. Psychol Assess. 2023 Jan;35(1):1-11. doi: 10.1037/pas0001183. Epub 2022 Sep 29. PMID 36174166
- [Background] Landry SH, Zucker TA, Williams JM, Merz EC, Guttentag CL, Taylor HB. Improving school readiness of high-risk preschoolers: Combining high quality instructional strategies with responsive training for teachers and parents. Early Childhood Research Quarterly. 2017;40:38-51.
- [Background] Landry SH, Taylor HB, Guttentag C, Smith KE. Responsive parenting: Closing the learning gap for children with early developmental problems. International review of research in mental retardation. 2008;36:27-60.
- [Background] Landry SH, Smith KE, Swank PR, Zucker T, Crawford AD, Solari EF. The effects of a responsive parenting intervention on parent-child interactions during shared book reading. Dev Psychol. 2012 Jul;48(4):969-86. doi: 10.1037/a0026400. Epub 2011 Nov 28. PMID 22122475
- [Background] Landry SH, Smith KE, Swank PR, Guttentag C. A responsive parenting intervention: the optimal timing across early childhood for impacting maternal behaviors and child outcomes. Dev Psychol. 2008 Sep;44(5):1335-53. doi: 10.1037/a0013030. PMID 18793067
- [Background] Krull KR, Hardy KK, Kahalley LS, Schuitema I, Kesler SR. Neurocognitive Outcomes and Interventions in Long-Term Survivors of Childhood Cancer. J Clin Oncol. 2018 Jul 20;36(21):2181-2189. doi: 10.1200/JCO.2017.76.4696. Epub 2018 Jun 6. PMID 29874137
- [Background] Kenney AE, Harman JL, Molnar AE Jr, Jurbergs N, Willard VW. Early Cognitive and Adaptive Functioning of Clinically Referred Infants and Toddlers with Cancer. J Clin Psychol Med Settings. 2020 Mar;27(1):41-47. doi: 10.1007/s10880-019-09619-1. PMID 30993575
- [Background] Kendall S, Bloomfield L. Developing and validating a tool to measure parenting self-efficacy. J Adv Nurs. 2005 Jul;51(2):174-81. doi: 10.1111/j.1365-2648.2005.03479.x. PMID 15963189
- [Background] Kaminski JW, Barrueco S, Kelleher KJ, Hoagwood K, Edwards A, Fox EG. Vital Signs for Pediatric Health: School Readiness. NAM Perspect. 2023 Jun 26;2023:10.31478/202306b. doi: 10.31478/202306b. eCollection 2023. No abstract available. PMID 37916064
- [Background] Vrijmoet-Wiersma CM, van Klink JM, Kolk AM, Koopman HM, Ball LM, Maarten Egeler R. Assessment of parental psychological stress in pediatric cancer: a review. J Pediatr Psychol. 2008 Aug;33(7):694-706. doi: 10.1093/jpepsy/jsn007. Epub 2008 Feb 19. PMID 18287109
- [Background] Jacola LM, Krull KR, Pui CH, Pei D, Cheng C, Reddick WE, Conklin HM. Longitudinal Assessment of Neurocognitive Outcomes in Survivors of Childhood Acute Lymphoblastic Leukemia Treated on a Contemporary Chemotherapy Protocol. J Clin Oncol. 2016 Apr 10;34(11):1239-47. doi: 10.1200/JCO.2015.64.3205. Epub 2016 Feb 8. PMID 26858334
- [Background] Hullmann SE, Wolfe-Christensen C, Meyer WH, McNall-Knapp RY, Mullins LL. The relationship between parental overprotection and health-related quality of life in pediatric cancer: the mediating role of perceived child vulnerability. Qual Life Res. 2010 Nov;19(9):1373-80. doi: 10.1007/s11136-010-9696-3. Epub 2010 Jun 24. PMID 20571917
- [Background] Hocking MC, McCurdy M, Turner E, Kazak AE, Noll RB, Phillips P, Barakat LP. Social competence in pediatric brain tumor survivors: application of a model from social neuroscience and developmental psychology. Pediatr Blood Cancer. 2015 Mar;62(3):375-84. doi: 10.1002/pbc.25300. Epub 2014 Nov 8. PMID 25382825
- [Background] Hile S, Erickson SJ, Agee B, Annett RD. Parental stress predicts functional outcome in pediatric cancer survivors. Psychooncology. 2014 Oct;23(10):1157-64. doi: 10.1002/pon.3543. Epub 2014 May 10. PMID 24817624
- [Background] Harman JL, Molnar AE Jr, Cox LE, Jurbergs N, Russell KM, Wise J, Willard VW. Parent-reported executive functioning in young children treated for cancer. Child Neuropsychol. 2019 May;25(4):548-560. doi: 10.1080/09297049.2018.1503647. Epub 2018 Jul 26. PMID 30049262
- [Background] Grieco JA, Evans CL, Yock TI, Pulsifer MB. Psychosocial and executive functioning late effects in pediatric brain tumor survivors after proton radiation. Childs Nerv Syst. 2024 Nov;40(11):3553-3561. doi: 10.1007/s00381-024-06579-2. Epub 2024 Sep 2. PMID 39222091
- [Background] Goodman R. The Strengths and Difficulties Questionnaire: a research note. J Child Psychol Psychiatry. 1997 Jul;38(5):581-6. doi: 10.1111/j.1469-7610.1997.tb01545.x. PMID 9255702
- [Background] Godoy PBG, Simionato NM, de Mello CB, Suchecki D. Assessment of Executive Functions after Treatment of Childhood Acute Lymphoid Leukemia: a Systematic Review. Neuropsychol Rev. 2020 Sep;30(3):386-406. doi: 10.1007/s11065-020-09446-4. Epub 2020 Jul 27. PMID 32720195
- [Background] French AE, Tsangaris E, Barrera M, Guger S, Brown R, Urbach S, Stephens D, Nathan PC. School attendance in childhood cancer survivors and their siblings. J Pediatr. 2013 Jan;162(1):160-5. doi: 10.1016/j.jpeds.2012.06.066. Epub 2012 Jul 24. PMID 22835883
- [Background] Fehr KK, Leraas BC, Littles MMD. Behavioral Health Needs, Barriers, and Parent Preferences in Rural Pediatric Primary Care. J Pediatr Psychol. 2020 Sep 1;45(8):910-920. doi: 10.1093/jpepsy/jsaa057. PMID 32766670
- [Background] Elling S, Lentz L, de Jong M, van den Bergh H. Measuring the quality of governmental websites in a controlled versus an online setting with the 'Website Evaluation Questionnaire'. Government Information Quarterly. 2012;29(3):383-93.
- [Background] Eisenberg N, Valiente C, Eggum ND. Self-Regulation and School Readiness. Early Educ Dev. 2010 Sep 1;21(5):681-698. doi: 10.1080/10409289.2010.497451. PMID 21234283
- [Background] Duncan GJ, Dowsett CJ, Claessens A, Magnuson K, Huston AC, Klebanov P, Pagani LS, Feinstein L, Engel M, Brooks-Gunn J, Sexton H, Duckworth K, Japel C. School readiness and later achievement. Dev Psychol. 2007 Nov;43(6):1428-1446. doi: 10.1037/0012-1649.43.6.1428. PMID 18020822
- [Background] Dumka, L. E., Stoerzinger, H. D., Jackson, K. M., & Roosa, M. W. (1996). Examination of the Cross-Cultural and Cross-Language Equivalence of the Parenting Self-Agency Measure. Family Relations, 45(2), 216-222. https://doi.org/10.2307/585293
- [Background] Denham SA. Social-Emotional Competence as Support for School Readiness: What Is It and How Do We Assess It? Early Education and Development. 2006;17(1):57-89. doi: 10.1207/s15566935eed1701_4
- [Background] Denham SA, Brown C. "Plays Nice With Others": Social-Emotional Learning and Academic Success. Early Education and Development. 2010;21(5):652-80. doi: 10.1080/10409289.2010.497450.
- [Background] Curtis ME, Clingan SE, Guo H, Zhu Y, Mooney LJ, Hser YI. Disparities in digital access among American rural and urban households and implications for telemedicine-based services. J Rural Health. 2022 Jun;38(3):512-518. doi: 10.1111/jrh.12614. Epub 2021 Aug 6. PMID 34355427
- [Background] Cox LE, Kenney AE, Harman JL, Jurbergs N, Molnar AE Jr, Willard VW. Psychosocial Functioning of Young Children Treated for Cancer: Findings From a Clinical Sample. J Pediatr Oncol Nurs. 2019 Jan/Feb;36(1):17-23. doi: 10.1177/1043454218813905. PMID 30798688
- [Background] Cortes Pascual A, Moyano Munoz N, Quilez Robres A. The Relationship Between Executive Functions and Academic Performance in Primary Education: Review and Meta-Analysis. Front Psychol. 2019 Jul 11;10:1582. doi: 10.3389/fpsyg.2019.01582. eCollection 2019. PMID 31354585
- [Background] Raj SP, Antonini TN, Oberjohn KS, Cassedy A, Makoroff KL, Wade SL. Web-Based Parenting Skills Program for Pediatric Traumatic Brain Injury Reduces Psychological Distress Among Lower-Income Parents. J Head Trauma Rehabil. 2015 Sep-Oct;30(5):347-56. doi: 10.1097/HTR.0000000000000052. PMID 24842588
- [Background] Campbell LK, Scaduto M, Van Slyke D, Niarhos F, Whitlock JA, Compas BE. Executive function, coping, and behavior in survivors of childhood acute lymphocytic leukemia. J Pediatr Psychol. 2009 Apr;34(3):317-27. doi: 10.1093/jpepsy/jsn080. Epub 2008 Jul 30. PMID 18667478
- [Background] Burek B, Ford MK, Hooper M, Green R, Kohut SA, Andrade BF, Ravi M, Sananes R, Desrocher M, Miller SP, Wade SL, Williams TS. Transdiagnostic feasibility trial of internet-based parenting intervention to reduce child behavioural difficulties associated with congenital and neonatal neurodevelopmental risk: introducing I-InTERACT-North. Clin Neuropsychol. 2021 Jul;35(5):1030-1052. doi: 10.1080/13854046.2020.1829071. Epub 2020 Oct 8. PMID 33028141
- [Background] Boterhoven de Haan KL, Hafekost J, Lawrence D, Sawyer MG, Zubrick SR. Reliability and validity of a short version of the general functioning subscale of the McMaster Family Assessment Device. Fam Process. 2015 Mar;54(1):116-23. doi: 10.1111/famp.12113. Epub 2014 Nov 11. PMID 25385473
- [Background] Bird M, Li L, Ouellette C, Hopkins K, McGillion MH, Carter N. Use of Synchronous Digital Health Technologies for the Care of Children With Special Health Care Needs and Their Families: Scoping Review. JMIR Pediatr Parent. 2019 Nov 21;2(2):e15106. doi: 10.2196/15106. PMID 31750840
- [Background] Beauchamp MH, Seguin M, Gagner C, Lalonde G, Bernier A. The PARENT model: a pathway approach for understanding parents' role after early childhood mild traumatic brain injury. Clin Neuropsychol. 2021 Jul;35(5):846-867. doi: 10.1080/13854046.2020.1834621. Epub 2020 Oct 26. PMID 33103594
- [Background] Baumel A, Fleming T, Schueller SM. Digital Micro Interventions for Behavioral and Mental Health Gains: Core Components and Conceptualization of Digital Micro Intervention Care. J Med Internet Res. 2020 Oct 29;22(10):e20631. doi: 10.2196/20631. PMID 33118946
- [Background] Aguilar JM, Cassedy AE, Shultz EL, Kirkwood MW, Stancin T, Yeates KO, Taylor HG, Wade SL. A Comparison of 2 Online Parent Skills Training Interventions for Early Childhood Brain Injury: Improvements in Internalizing and Executive Function Behaviors. J Head Trauma Rehabil. 2019 Mar/Apr;34(2):65-76. doi: 10.1097/HTR.0000000000000443. PMID 30499926
- [Background] Ackerman DJ, Friedman-Krauss AH. Preschoolers' executive function: Importance, contributors, research needs and assessment options. ETS Research Report Series. 2017;2017(1):1-24.
- [Background] Ach E, Gerhardt CA, Barrera M, Kupst MJ, Meyer EA, Patenaude AF, Vannatta K. Family factors associated with academic achievement deficits in pediatric brain tumor survivors. Psychooncology. 2013 Aug;22(8):1731-7. doi: 10.1002/pon.3202. Epub 2012 Oct 12. PMID 23059621